CLINICAL TRIAL: NCT03706157
Title: Kinectics of Distribution of Doxorubicin-Lipiodol Emulsion in c-TACE: a Pilot Study
Brief Title: Kinectics of Distribution of Doxorubicin-Lipiodol Emulsion in c-TACE
Acronym: CineDoxo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 7040
Record Dates: First submitted 2018-10-02; First posted 2018-10-15 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2019-08

CONDITIONS: Hepato Cellular Carcinoma
Keywords: Conventional transarterial chemoembolization (c-TACE); Doxorubicin; Kinetics of distribution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodinate contrast (Active Comparator): Doxorubicin solution reconstituted in 5 mL iso-osmolar ionic iodinated contrast media
  Interventions: Drug: Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc iso-osmolar ionic iodinated contrast media
- Normal saline (Active Comparator): Doxorubicin solution reconstituted in 5 mL normal saline
  Interventions: Drug: Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc normal saline

INTERVENTIONS:
Drug: Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc iso-osmolar ionic iodinated contrast media — Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc iso-osmolar ionic iodinated contrast media
  Arms: Iodinate contrast
Drug: Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc normal saline — Super selective transarterial chemoembolization of CHC, with doxorubicin reconstituted in 5cc normal saline
  Arms: Normal saline

SUMMARY:
Conventional transarterial chemoembolization with Doxorubicin (c-TACE) is the gold standard treatment for Hepato Cellular Carcinoma (HCC) stage B (BCLC) / stages A and B (Child-Pugh). Clinical recommendations for cTACE indicate that the doxorubicin solution may be reconstituted in either aqueous solution or iso-osmolar ionic iodinated contrast media. There is no consensus on which solvent should be used. Hence, the clinical evaluation of Lipiodol cTACE would benefit from a standardization in the reconstitution of the drug. In this study, the comparison of the kinetics of distribution of the drug within the tumor micro-environment is expected to allow for comparison of drug solvents.

This pilot study aims at evaluating the kinetics of distribution of the drug within the tumor micro-environment, for the two main solvents used in reconstituting the drug, namely normal saline and contrast media. The kinetics of distribution in the tumor will be evaluated primarily through regular biopsy sampling, and secondary with confocal laser endomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18)
* Informed consent
* CHC Child-Pugh stage A or B, BCLC stage B
* Referred for chemoembolization of a non-surgery-candidate CHC
* Blood test results compatible with cTACE (INR ≤ 1,5, ASAT/ALAT<5N, albumine>2,5g/dl)

Exclusion Criteria:

* Contraindication to cTACE, angiography, confocal laser endomicroscopy or liver biopsy Hyperthyroidism
* Contraindication to the use of fluorescein, Ariblastine,Lipiodol, Visipaque, Gelita spon, Avitene
* extra hepatic metastasis
* Subcapsular or exophytic tumor impeding direct percutaneous access through healthy liver tissue
* Waiting list for liver transplant
* Complete portal venous thrombosis or flow inversion
* Pregnancy or breast feeding
* Protected major (Guardianship)
* Patient in situation of exclusion (determined by a previous or ongoing study)
* Subject incapacity to understand informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Histological analysis of biopsy samples for the evaluation of the kinetics of distribution of doxorubicine in tumor compartments depending on the solvent used for drug reconstitution | T0: 1 min before cTACE drug injection star
  Biopsy samples of liver tumor tissue. Histological analysis will provide a quantification of the doxorubicin drug in tumor compartment.
Histological analysis of biopsy samples for the evaluation of the kinetics of distribution of doxorubicine in tumor compartments depending on the solvent used for drug reconstitution | T1 : 2 min after cTACE drug injection started
  Biopsy samples of liver tumor tissue. Histological analysis will provide a quantification of the doxorubicin drug in tumor compartment.
Histological analysis of biopsy samples for the evaluation of the kinetics of distribution of doxorubicine in tumor compartments depending on the solvent used for drug reconstitution | T2: 1 second after half of cTACE drug has been injected
  Biopsy samples of liver tumor tissue. Histological analysis will provide a quantification of the doxorubicin drug in tumor compartment.
Histological analysis of biopsy samples for the evaluation of the kinetics of distribution of doxorubicine in tumor compartments depending on the solvent used for drug reconstitution | T3: 1 min after cTACE drug injection is completed
  Biopsy samples of liver tumor tissue. Histological analysis will provide a quantification of the doxorubicin drug in tumor compartment.

SECONDARY OUTCOMES:
In vivo evaluation of the kinetics of distribution of doxorubicine in tumoral tissue with confocal laser endomicroscopy, depending on the solvent used for drug reconstitution | 1 min before cTACE drug injection starts,
  Continuous image recording (videos) through the course of the cTACE drug injection, from 1 minute before drug injection starts to the time when cTACE drug injection is completed
In vivo evaluation of the kinetics of distribution of doxorubicine in tumoral tissue with confocal laser endomicroscopy, depending on the solvent used for drug reconstitution | 2 min after cTACE drug injection started,
  Continuous image recording (videos) through the course of the cTACE drug injection, from 1 minute before drug injection starts to the time when cTACE drug injection is completed
In vivo evaluation of the kinetics of distribution of doxorubicine in tumoral tissue with confocal laser endomicroscopy, depending on the solvent used for drug reconstitution | 1 second after half of cTACE drug has been injected,
  Continuous image recording (videos) through the course of the cTACE drug injection, from 1 minute before drug injection starts to the time when cTACE drug injection is completed
In vivo evaluation of the kinetics of distribution of doxorubicine in tumoral tissue with confocal laser endomicroscopy, depending on the solvent used for drug reconstitution | 1 min after cTACE drug injection is completed,
  Continuous image recording (videos) through the course of the cTACE drug injection, from 1 minute before drug injection starts to the time when cTACE drug injection is completed

CONTACTS AND LOCATIONS:
Overall Officials: Iuian 03 69 55 15 27, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France